CLINICAL TRIAL: NCT03418454
Title: The Oral Microbiome as a Prognostic Tool in Oral Malignant and Premalignant Lesions and in Medication Related Osteonecrosis of the Jaw
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Irit Allon, DMD, PhD, Principal Investigator, Barzilai Medical Center
Other Study IDs: BRZ 0062-17 CTIL
Record Dates: First submitted 2018-01-16; First posted 2018-02-01 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Oral Squamous Cell Carcinoma; Medication Related Osteonecrosis of the Jaw; Oral Epithelial Dysplasia
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Oral Squamous Cell Carcinoma: Buccal mucosa samples for Extraction of BACTERIAL DNA
  Interventions: Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA
- Oral Epithelial Dysplasia: Buccal mucosa samples for Extraction of BACTERIAL DNA
  Interventions: Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA
- Control: Healthy age matched patients: Buccal mucosa samples for Extraction of BACTERIAL DNA
  Interventions: Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA
- Osteonecrosis of the Jaw: Buccal mucosa samples for Extraction of BACTERIAL DNA
  Interventions: Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA
- Underlying disease, no necrosis of the jaw: Buccal mucosa samples for Extraction of BACTERIAL DNA
  Interventions: Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA

INTERVENTIONS:
Diagnostic Test: Buccal mucosa samples for Extraction of BACTERIAL DNA — Sampling of the buccal mucosa after informed consent and prior to routine treatment. Similar sampling on follow up after 3,6,9,12 months.
  Extracted BACTERIAL DNA (and not human DNA) from clinical samples will be sequenced and analyzed for the 16s rRNA (BACTERIAL ribosome).

SUMMARY:
Oral squamous cell carcinoma (OSCC) is the most common malignant tumor of the head and neck, and its incidence has increased in recent years. Extensive surgery with neck dissection and chemo/radio/ targeted therapy is the current treatment for OSCC, and despite great progress in chemotherapy, radiotherapy, and targeted therapy in the last three decades, the prognosis of OSCC is still poor due to aggressive local invasion and metastasis, which lead to recurrence. Postoperative tumor recurrence confers a poor prognosis in OSCC and a poor quality of life. The 5-year survival rate is over 90% in OSCC patients without recurrence and 30% in patients with recurrence, with a median survival of 76.8 months in patients without recurrence and 42.5 months in patients with recurrence . Therefore, it is important to identify biomarkers that may predict the postoperative recurrence of OSCC. Also, some of the OSCC are preceded by precursor lesions. In the oral cavity the most common lesions recognized as potentially malignant are leukoplakia and erythroplakia, but it is also apparent that as many as 50% of OSCC arise from apparently clinically normal mucosa. The prognostic significance of an individual lesion is difficult to determine. At present therefore, the gold standard for the assessment of oral potentially malignant lesions is microscopic evaluation of haematoxylin and eosin stained sections for the presence of architectural and cytological changes, which are generally referred to as oral epithelial dysplasia (OED). The human microbiome is defined as the collective genomes of the microbes (composed of bacteria, bacteriophages, fungi, protozoa and viruses) that live inside and on the human body, and there are approximately 10 microbes and 100 microbial genes for each human cell and gene respectively. With the advent of next generation sequencing technology, the Human Microbiome Project delineated the composition of healthy microbial communities associated to different body sites in healthy individuals, including the oral cavity [Human microbiome consortium]. As opposed to a normal (healthy) microbiome, a disrupted microbiome or dysbiosis represents the lack of equilibrium, and is hypothetically related to disease. Interestingly, the healthy oral microbiome shows relative intraindividual stability over time, suggesting that differences in microbiome profiles may serve as useful tools for the identification of disease states. The working hypothesis is that in OSCC patients, the oral microbiome is altered in comparison to healthy individuals and certain microbial signatures are characteristic of healthy versus disease. In addition, in precursor conditions, i.e., oral epithelial dysplasia (OED), a partial alteration in the composition of the microbiome may predict the progression to malignancy.Also, during treatment, it could be that specific microbial signatures are associated with incomplete eradication, tendency to local recurrence or metastatic potential.Correlations to local recurrence (LR), distant metastases (DM) or disease free survival (DFS) adjusted to clinicopathologic correlations will be sought. In this study, buccal mucosa samples will be collected from patients with OSCC, OED and from healthy individuals , after signing for informed consent, according to Helsinki protocol. Routine pathologic diagnosis will be performed by expert Pathology physicians in our center. Data will be correlated to demographic and clinical data obtained from medical records. This will be carried out in line with institutional ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients biopsied with OSCC
* Patients biopsied with oral premalignant lesions
* Patients biopsied with osteonecrosis of the jaw
* healthy age matched patients that visit the oral and maxillofacial clinic for other purposes such as extraction, reactive lesions

Exclusion Criteria:

* Patients receiving antimicrobial treatment in the previous 3 months
* Patients receiving radiotherapy
* Patients receiving chemo/immunotherapy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the Oral & Maxillofacial Surgery outpatient Clinique at the Barzilai Medical Center, Ashkelon, Israel
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome characterization day 1 of the study | Day 1 of each participant
  Extracted BACTERIAL DNA sequenced by amplification of the V4 region of 16s rRNA (BACTERIAL ribosome). The samples will be obtained by buccal mucosa swabs from all subjects at the clinic visit (day 1). FLOQ swabs (Copan) will be rubbed on the inner cheek mucosa that looks macroscopically normal. The swab will be immediately placed in a 15ml polypropylene tube containing 1 ml of Molecular grade PBS. Samples will be kept at 4oC until frozen at -80oC. Each sample will be assigned a protocol serial number, de-identified from the subject.
Microbiome characterization month 3 of the study | Month 3 of each participant
  1Extracted BACTERIAL DNA sequenced by amplification of the V4 region of 16s rRNA (BACTERIAL ribosome). The samples will be obtained by buccal mucosa swabs from all subjects at the clinic visit (month 3). FLOQ swabs (Copan) will be rubbed on the inner cheek mucosa that looks macroscopically normal. The swab will be immediately placed in a 15ml polypropylene tube containing 1 ml of Molecular grade PBS. Samples will be kept at 4oC until frozen at -80oC. Each sample will be assigned a protocol serial number, de-identified from the subject.
Microbiome characterization month 6 of the study | Month 6 of each participant
  Extracted BACTERIAL DNA sequenced by amplification of the V4 region of 16s rRNA (BACTERIAL ribosome). The samples will be obtained by buccal mucosa swabs from all subjects at the clinic visit (month 6). FLOQ swabs (Copan) will be rubbed on the inner cheek mucosa that looks macroscopically normal. The swab will be immediately placed in a 15ml polypropylene tube containing 1 ml of Molecular grade PBS. Samples will be kept at 4oC until frozen at -80oC. Each sample will be assigned a protocol serial number, de-identified from the subject.
Microbiome characterization month 9 of the study | Month 9 of each participant
  Extracted BACTERIAL DNA sequenced by amplification of the V4 region of 16s rRNA (BACTERIAL ribosome). The samples will be obtained by buccal mucosa swabs from all subjects at the clinic visit (month 9). FLOQ swabs (Copan) will be rubbed on the inner cheek mucosa that looks macroscopically normal. The swab will be immediately placed in a 15ml polypropylene tube containing 1 ml of Molecular grade PBS. Samples will be kept at 4oC until frozen at -80oC. Each sample will be assigned a protocol serial number, de-identified from the subject.
Microbiome characterization month 12 of the study | Month 12 of each participant
  3. Extracted BACTERIAL DNA sequenced by amplification of the V4 region of 16s rRNA (BACTERIAL ribosome). The samples will be obtained by buccal mucosa swabs from all subjects at the clinic visit (month 12). FLOQ swabs (Copan) will be rubbed on the inner cheek mucosa that looks macroscopically normal. The swab will be immediately placed in a 15ml polypropylene tube containing 1 ml of Molecular grade PBS. Samples will be kept at 4oC until frozen at -80oC. Each sample will be assigned a protocol serial number, de-identified from the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bagan JV, Scully C. Recent advances in Oral Oncology 2007: epidemiology, aetiopathogenesis, diagnosis and prognostication. Oral Oncol. 2008 Feb;44(2):103-8. doi: 10.1016/j.oraloncology.2008.01.008. PMID 18252251
- [Background] Camisasca DR, Silami MA, Honorato J, Dias FL, de Faria PA, Lourenco Sde Q. Oral squamous cell carcinoma: clinicopathological features in patients with and without recurrence. ORL J Otorhinolaryngol Relat Spec. 2011;73(3):170-6. doi: 10.1159/000328340. Epub 2011 May 27. PMID 21625192
- [Background] Lindenblatt Rde C, Martinez GL, Silva LE, Faria PS, Camisasca DR, Lourenco Sde Q. Oral squamous cell carcinoma grading systems--analysis of the best survival predictor. J Oral Pathol Med. 2012 Jan;41(1):34-9. doi: 10.1111/j.1600-0714.2011.01068.x. Epub 2011 Sep 8. PMID 21902722
- [Background] Dietert RR, Silbergeld EK. Biomarkers for the 21st century: listening to the microbiome. Toxicol Sci. 2015 Apr;144(2):208-16. doi: 10.1093/toxsci/kfv013. Epub 2015 Mar 20. PMID 25795652
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Li K, Bihan M, Yooseph S, Methe BA. Analyses of the microbial diversity across the human microbiome. PLoS One. 2012;7(6):e32118. doi: 10.1371/journal.pone.0032118. Epub 2012 Jun 13. PMID 22719823
- [Background] Ding T, Schloss PD. Dynamics and associations of microbial community types across the human body. Nature. 2014 May 15;509(7500):357-60. doi: 10.1038/nature13178. Epub 2014 Apr 16. PMID 24739969
- [Background] Meyer MS, Joshipura K, Giovannucci E, Michaud DS. A review of the relationship between tooth loss, periodontal disease, and cancer. Cancer Causes Control. 2008 Nov;19(9):895-907. doi: 10.1007/s10552-008-9163-4. Epub 2008 May 14. PMID 18478344
- [Background] Fitzpatrick SG, Katz J. The association between periodontal disease and cancer: a review of the literature. J Dent. 2010 Feb;38(2):83-95. doi: 10.1016/j.jdent.2009.10.007. Epub 2009 Nov 4. PMID 19895866
- [Background] Ahn J, Segers S, Hayes RB. Periodontal disease, Porphyromonas gingivalis serum antibody levels and orodigestive cancer mortality. Carcinogenesis. 2012 May;33(5):1055-8. doi: 10.1093/carcin/bgs112. Epub 2012 Feb 26. PMID 22367402
- [Background] Yu G, Gail MH, Shi J, Klepac-Ceraj V, Paster BJ, Dye BA, Wang GQ, Wei WQ, Fan JH, Qiao YL, Dawsey SM, Freedman ND, Abnet CC. Association between upper digestive tract microbiota and cancer-predisposing states in the esophagus and stomach. Cancer Epidemiol Biomarkers Prev. 2014 May;23(5):735-41. doi: 10.1158/1055-9965.EPI-13-0855. Epub 2014 Apr 3. PMID 24700175
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Meurman JH, Uittamo J. Oral micro-organisms in the etiology of cancer. Acta Odontol Scand. 2008;66(6):321-6. doi: 10.1080/00016350802446527. PMID 18821087
- [Background] Meurman JH. Oral microbiota and cancer. J Oral Microbiol. 2010 Aug 10;2. doi: 10.3402/jom.v2i0.5195. PMID 21523227
- [Background] Nagy KN, Sonkodi I, Szoke I, Nagy E, Newman HN. The microflora associated with human oral carcinomas. Oral Oncol. 1998 Jul;34(4):304-8. PMID 9813727
- [Background] Pushalkar S, Ji X, Li Y, Estilo C, Yegnanarayana R, Singh B, Li X, Saxena D. Comparison of oral microbiota in tumor and non-tumor tissues of patients with oral squamous cell carcinoma. BMC Microbiol. 2012 Jul 20;12:144. doi: 10.1186/1471-2180-12-144. PMID 22817758
- [Background] Schmidt BL, Kuczynski J, Bhattacharya A, Huey B, Corby PM, Queiroz EL, Nightingale K, Kerr AR, DeLacure MD, Veeramachaneni R, Olshen AB, Albertson DG. Changes in abundance of oral microbiota associated with oral cancer. PLoS One. 2014 Jun 2;9(6):e98741. doi: 10.1371/journal.pone.0098741. eCollection 2014. PMID 24887397
- [Background] Ahn J, Chen CY, Hayes RB. Oral microbiome and oral and gastrointestinal cancer risk. Cancer Causes Control. 2012 Mar;23(3):399-404. doi: 10.1007/s10552-011-9892-7. Epub 2012 Jan 22. PMID 22271008
- [Background] Guerrero-Preston R, Godoy-Vitorino F, Jedlicka A, Rodriguez-Hilario A, Gonzalez H, Bondy J, Lawson F, Folawiyo O, Michailidi C, Dziedzic A, Thangavel R, Hadar T, Noordhuis MG, Westra W, Koch W, Sidransky D. 16S rRNA amplicon sequencing identifies microbiota associated with oral cancer, human papilloma virus infection and surgical treatment. Oncotarget. 2016 Aug 9;7(32):51320-51334. doi: 10.18632/oncotarget.9710. PMID 27259999
- [Background] Speight PM. Update on oral epithelial dysplasia and progression to cancer. Head Neck Pathol. 2007 Sep;1(1):61-6. doi: 10.1007/s12105-007-0014-5. Epub 2007 Nov 30. No abstract available. PMID 20614284
- [Background] Sedghizadeh PP, Yooseph S, Fadrosh DW, Zeigler-Allen L, Thiagarajan M, Salek H, Farahnik F, Williamson SJ. Metagenomic investigation of microbes and viruses in patients with jaw osteonecrosis associated with bisphosphonate therapy. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Dec;114(6):764-70. doi: 10.1016/j.oooo.2012.08.444. PMID 23159114
- [Background] Kolenbrander PE, Andersen RN, Blehert DS, Egland PG, Foster JS, Palmer RJ Jr. Communication among oral bacteria. Microbiol Mol Biol Rev. 2002 Sep;66(3):486-505, table of contents. doi: 10.1128/MMBR.66.3.486-505.2002. PMID 12209001
- [Background] Ribeiro GH, Chrun ES, Dutra KL, Daniel FI, Grando LJ. Osteonecrosis of the jaws: a review and update in etiology and treatment. Braz J Otorhinolaryngol. 2017 Jun 24;84(1):102-8. doi: 10.1016/j.bjorl.2017.05.008. Online ahead of print. PMID 28712852
- [Background] Voss PJ, Poxleitner P, Schmelzeisen R, Stricker A, Semper-Hogg W. Update MRONJ and perspectives of its treatment. J Stomatol Oral Maxillofac Surg. 2017 Sep;118(4):232-235. doi: 10.1016/j.jormas.2017.06.012. Epub 2017 Jul 8. PMID 28697987